CLINICAL TRIAL: NCT02583451
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, 4-Period Crossover Study to Evaluate the Effect of Lemborexant Versus Placebo on Driving Performance in Healthy Adult and Elderly Subjects
Brief Title: Study to Evaluate the Effect of Lemborexant Versus Placebo on Driving Performance in Healthy Adult and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: E2006-E044-106
Record Dates: First submitted 2015-10-16; First posted 2015-10-22 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy Participants
MeSH Terms: interventions — zopiclone; lemborexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A (Experimental): Treatment A is a placebo tablet matching lemborexant and placebo tablet matching zopiclone on nights in the clinic; placebo tablet matching lemborexant on nights at home.
  Interventions: Drug: Placebo tablet matching lemborexant; Drug: Placebo tablet matching zopiclone
- Treatment B (Experimental): Treatment B is zopiclone 7.5 mg tablet and placebo tablet matching lemborexant on nights in the clinic; placebo tablet matching lemborexant on nights at home.
  Interventions: Drug: Placebo tablet matching lemborexant; Drug: Zopiclone 7.5 mg
- Treatment C (Experimental): Treatment C is lemborexant 2.5 mg tablet and placebo tablet matching zopiclone on nights in the clinic; lemborexant 2.5 mg tablet on nights at home.
  Interventions: Drug: Placebo tablet matching zopiclone; Drug: Lemborexant 2.5 mg
- Treatment D (Experimental): Treatment D is lemborexant 5 mg tablet and placebo tablet matching zopiclone on nights in the clinic; lemborexant 5 mg tablet on nights at home.
  Interventions: Drug: Placebo tablet matching zopiclone; Drug: Lemborexant 5 mg
- Treatment E (Experimental): Treatment E is lemborexant 10 mg tablet and placebo tablet matching zopiclone on nights in the clinic; lemborexant 10 mg tablet on nights at home.
  Interventions: Drug: Placebo tablet matching zopiclone; Drug: Lemborexant 10 mg

INTERVENTIONS:
Drug: Placebo tablet matching lemborexant — Tablet form taken orally at bedtime.
  Arms: Treatment A; Treatment B
Drug: Placebo tablet matching zopiclone — Tablet form taken orally at bedtime.
  Arms: Treatment A; Treatment C; Treatment D; Treatment E
Drug: Zopiclone 7.5 mg — 7.5 mg tablet taken orally at bedtime.
  Arms: Treatment B
Drug: Lemborexant 2.5 mg — 2.5 tablet taken orally at bedtime.
  Arms: Treatment C
Drug: Lemborexant 5 mg — 5 mg tablet taken orally at bedtime.
  Arms: Treatment D
Drug: Lemborexant 10 mg — 10 mg tablet taken orally at bedtime.
  Arms: Treatment E

SUMMARY:
This is a randomized, double-blind, placebo- and active-controlled, 4-period crossover study of lemborexant in healthy adult and elderly subjects to evaluate driving performance

DETAILED DESCRIPTION:
The study will have 2 phases, Prerandomization and Randomization. The Prerandomization Phase will consist of 2 periods that will last up to a maximum of 21 days: Screening and Baseline. The Randomization Phase will comprise of four, 9-day treatment periods (Treatment Period 1 - Treatment Period 4) with a minimum 14-day washout between treatment periods, and a follow-up interval of at least 14 days after Treatment Period 4 before the end-of-study (EOS) visit. Participants will be randomized to 1 of 12 sequences in an incomplete blocks design.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female, aged 21 years or older at Screening
2. Regular time spent in bed between 7.0 and 8.5 hours per night
3. Regular bedtime, defined as the time the participant attempts to fall asleep, between 22:00 hours and 01:00 hours, and regular waketime, defined as the time the participant gets out of bed for the day, between 05:00 hours and 09:00 hours
4. Body mass index (BMI) ≥18 and <31 kg/m2 at Screening
5. Subjective sleep onset latency (sSOL) <30 minutes and subjective wake after sleep onset (sWASO) <60 minutes on the Sleep Diary
6. At least 3 years of experience driving at least 3000 km per year
7. Holds a valid license to drive a vehicle in the European Union (EU) as confirmed at the Screening visit
8. Has driving ability during the practice driving test that is judged to be adequate by the driving instructor
9. Able to communicate adequately (written and verbal) in either Dutch or English as determined by the investigator

Exclusion Criteria:

1. A current complaint or diagnosis of insomnia disorder (per either The Diagnostic and Statistical Manual of Mental Disorders Version IV [DSM-IV] or Version 5 [DSM-5] criteria), sleep-related breathing disorder, periodic limb movement disorder, restless legs or narcolepsy, or an exclusionary score on a subscale of the SLEEP50
2. Habitually naps more than 3 times per week
3. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of B-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
4. Females of childbearing potential who:

   * Had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period or for 28 days after study drug discontinuation.
   * Are currently abstinent, and do not agree to use a double-barrier method (as described above) or refrain from sexually active during the study period or for 28 days after study drug discontinuation.
   * Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study or for 28 days after study drug discontinuation. (NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing]).
5. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception throughout the study period or for 28 days after study drug discontinuation). No sperm donation is allowed during the study period or for 28 days after study drug discontinuation.
6. Clinically significant illness that requires medical treatment between Screening and Baseline
7. Any clinically abnormal symptom or organ impairment found by medical history at Screening or Baseline and physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment
8. Has a QT interval corrected using Fridericia's formula interval (QTcF interval) >450 ms demonstrated on repeated ECGs (repeated only if initial ECG showed corrected QT interval (QTc) >450 ms) at Screening or Baseline
9. Has a history of or a family history of congenital QT prolongation or with a history of risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome), or uses concomitant medications that prolong the QT/QT interval corrected for heart rate (QTc interval)
10. Has systolic blood pressure (BP) >140 mmHg (age 21-59) or >150 mmHg (age ≥60) or diastolic BP >90 mmHg (all ages) at Screening or Baseline
11. Has a resting heart rate <50 or ≥100 beats/min at Screening or Baseline
12. Has a history of drug or alcohol dependency or abuse (as defined by DSM-5 criteria) within approximately 2 years before Screening
13. Any suicidal ideation with intent with or without a plan within 6 months of the Screening Period (ie, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the C-SSRS)
14. Habitually consumes more than 14 drinks per week (females) or more than 21 drinks per week (males)
15. Has a positive alcohol breathalyzer test at Screening or Baseline check-in
16. Smokes more than 6 cigarettes per day habitually and is unwilling to abstain from smoking cigarettes on evenings spent in the clinic until discharge after the driving test
17. Habitually consumes more than 3 cups of caffeinated beverages per day
18. Used any prohibited prescription or over-the-counter (OTC) concomitant medications within 1 week prior to starting the Sleep Diary during the Screening Period
19. Transmeridian travel across more than 3 time zones in the 2 weeks before Screening, or between Screening and Baseline or plans for transmeridian travel across more than 3 time zones during the study
20. A positive urine drug test at Screening or unwilling to refrain from use of illegal recreational drugs or marijuana during the study
21. Hypersensitivity to the study drug or any of the excipients or to zopiclone
22. Participated (received investigational product) in another clinical trial less than 1 month (or 5 elimination half-lives of the investigational product) before dosing or is currently enrolled in another clinical study

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change of standard deviation of lateral position (SDLP) during an on-road driving test | Day 2, Day 9, Day 23, Day 30, Day 44, Day 51, Day 65, and Day 72

SECONDARY OUTCOMES:
Number of lapses on the driving test | Day 2, Day 9, Day 23, Day 30, Day 44, Day 51, Day 65, and Day 72
Outliers on SDLP | Day 2, Day 9, Day 23, Day 30, Day 44, Day 51, Day 65, and Day 72
Outliers on number of lapses | Day 2, Day 9, Day 23, Day 30, Day 44, Day 51, Day 65, and Day 72
Percentage of participants who never started a scheduled driving test or who stopped prematurely | Day 2, Day 9, Day 23, Day 30, Day 44, Day 51, Day 65, and Day 72
Standard deviation of lateral position (SDLP) during an on-road driving test, by age group | Day 2, Day 9, Day 23, Day 30, Day 44, Day 51, Day 65, and Day 72
Plasma concentration of lemborexant | Day 2, Day 9, Day 23, Day 30, Day 44, Day 51, Day 65, and Day 72
Number of lapses on the driving test, by age group | Day 2, Day 9, Day 23, Day 30, Day 44, Day 51, Day 65, and Day 72
Plasma concentration of S-zopiclone | Day 2, Day 9, Day 23, Day 30, Day 44, Day 51, Day 65, and Day 72

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Gotfried MH, Auerbach SH, Dang-Vu TT, Mishima K, Kumar D, Moline M, Malhotra M. Efficacy and safety of insomnia treatment with lemborexant in older adults: analyses from three clinical trials. Drugs Aging. 2024 Sep;41(9):741-752. doi: 10.1007/s40266-024-01135-8. Epub 2024 Aug 9. PMID 39120786
- [Derived] Vermeeren A, Jongen S, Murphy P, Moline M, Filippov G, Pinner K, Perdomo C, Landry I, Majid O, Van Oers ACM, Van Leeuwen CJ, Ramaekers JG, Vuurman EFPM. On-the-road driving performance the morning after bedtime administration of lemborexant in healthy adult and elderly volunteers. Sleep. 2019 Apr 1;42(4):zsy260. doi: 10.1093/sleep/zsy260. PMID 30597112